CLINICAL TRIAL: NCT05360589
Title: Assessment of Central and Peripheral Sensitization, and Pain Contributing Factors in Patients With Non-specific Shoulder Pain. A Case-control Study
Brief Title: Central and Peripheral Sensitization, and Pain Contributing Factors in Shoulder Pain Patients and Healthy People
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Collaborators: Centro Medico Albese (Unknown)
Responsible Party: Principal Investigator, Giacomo Carta, Principal Investigator, University of Turin, Italy
Other Study IDs: 7757/2022
Record Dates: First submitted 2022-04-14; First posted 2022-05-04 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; Central sensistization; Peripheral sensitization; Modulating factors; ICF; Disability
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shoulder non-specific pain: 68 adult gender-balanced subjects will be enrolled, reporting unilateral, atraumatic, and non-specific shoulder pain68 healthy subjects who regularly perform sports activities (at least one weekly session).
- Controls: 68 healthy subjects who regularly perform sports activities (at least one time/week) without shoulder pain will be recruited.

SUMMARY:
Compared to healthy subjects, central and peripheral sensitization will be investigated in patients with non-specific shoulder pain, since no data is available at the moment. The Central Sensitization Inventory (CSI) will be administered to assess sensitization in patients and controls, and changes in the mechanosensitivity of the upper limb will be assessed by checking for mechanical allodynia, hyperalgesia, and wind-up related to peripheral sensitization. Chronic pain mediators factors such as anxiety, depression, catastrophization, self-efficacy, and kinesiophobia will be investigated through validated rating scales. The Vagus Nerve neurodynamic test (VN-NDT) will be performed to assess any HR variability reduction related to stress mechanisms typical of chronic pain conditions. Finally, to health status of participants, following the biopsychosocial model, the Generic Core Set of the International Classification of the Functioning of Disability and Health (ICF) will be assessed.

DETAILED DESCRIPTION:
Introduction: Growing evidence shows that non-specific shoulder pain is a common musculoskeletal condition. It often involves a severe reduction in the functionality of the upper limb with a remarkable impact on daily life activities and social participation. Like back pain disorders, it is known that it has a high risk of chronification and is associated with central and peripheral sensitization phenomena. These processes are clinically detectable as hyperalgesia, allodynia, and wind-up phenomenon, but it is not yet explored if those processes are reported in shoulder pain patients. Moreover, modern clinical neuroscience had revealed that behavioral factors such as anxiety, depression, poor self-efficacy, kinesiphobia, and catastrophization contributes to pain chronification but a clear involvement of these factors has not been defined yet for shoulder pain. Considering that the relation between anatomical alterations detectable with imaging techniques is very poor when assessing chronic pain patients it is useful to explore this condition from a biopsychosocial point of view that nowadays is lacking.

To better define and treat non-specific shoulder pain patients, exploring central and peripheral sensitization, chronic pain contributing factors, and their health status is of paramount importance. Methods: A case-control study will be performed. Based on the best evidence the sample size was calculated. It was estimated 68 people with non-specific shoulder pain and 68 healthy controls are needed to be evaluated. All participants will fulfill the following validated rating scales exploring central sensitization, pain chronification factors, disability and health status. The disability will be assessed using The Shoulder Pain and Disability Index, central sensitization using the Central Sensitization Inventory (CSI), catastrophization using the Pain Catastrophizing Scale (PCS), kinesiophobia using the Tampa Scale for Kinesiophobia (TSK), anxiety and depression using the Hospital Anxiety Depression Scale (HADS) and self-efficacy using the Pain Self-efficacy Questionnaire (PSEQ). A trained physiotherapist will complete the ICF Generic Core Set, and after sharing it with the patient, a patient-clinician evaluation of the health status will be defined. Moreover, a clinical examination will be carried out to detect tactile and mechanical allodynia, wind-up phenomenon, and mechanosensitivity changes in the shoulder. A multivariate model will be considered for the statistical analysis to check for any confounding, and tests for estimating variance differences will be used.

Expected results: The study is expected to describe the relevance of processes related to central and peripheral sensitization in chronic shoulder pain patients, with a plausible difference between healthy controls. It will be possible to define the relevance of pain chronification factors and health status considering the complexity of pain from a biopsychosocial point of view. The investigators expect to identify which factors are related to disability and loss of participation in shoulder pain. Conclusion: The study is aimed to offer a multifactorial overview of patients with non-specific shoulder pain to provide tailored and precise rehabilitation programs, considering the clinical relevant factors and reducing the resource waste in less effective interventions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects giving their written consent to be enrolled in the study.
* Subjects aged more than 18 years old.
* Subjects reporting unilateral, atraumatic, and non-specific shoulder pain and/or mechanosensitivity changes in the shoulder region such as burning pain, shocks, and tingling pain.

Exclusion Criteria:

* Subjects presenting massive lesions, fractures, joint instability following dislocations or subluxations of the shoulder.
* Subjects presenting nerve conduction deficiency
* Subjects underwent at least once in their life shoulder prostheses and/or interventions that have altered the shoulder anatomy
* Subjects undergone shoulder surgery less than 2 years before the assessment.
* Subjects reporting a history of trauma and/or dislocation less than a year before the assessment.
* Subjects presenting central neurological diseases, neurodegenerative diseases, demyelinating acute diseases (ex: Guillane Barrè), oncology and psychiatry diseases, and diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with non-specific shoulder pain and healthy subjects that give their consent to be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Italian Central Sensitization Inventory (CSI-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be adopted to assess central sensitization. It consists of two sections. Part A is made up of 25 self-reported items, each rated on a scale from 0 to 5 (0=never and 4=always), for a maximum score of 100. Part B analyses the presence of commonly related symptoms. A total score < 40 shows good sensitivity to exclude the presence of signs and symptoms related to central sensitization.
Numeric Pain Rating Scale | The scale will be administered to assess the pain intensity during provocative tests during the clinical examination (day 1)
  pain intensity will be tested asking the standardized question " on a scale from 0 to 10 when 0 is no pain and 10 is the worst pain ever rate the pain intensity you feel in this moment in the body part assessed"
Quantitative sensory testing (QST) -Tactile discrimination | The outcome will be measured on day 1 for each site, by a physiotherapist during the clinical examination
  These tests will be adopted to assess peripheral and central sensitiazion phenomena. Tests will be administered once for each site, by a physiotherapist using Neuropen.
  -Tactile discrimination will be tested by administering an alternation of three tactile stimuli and three puncture stimuli at the level of the coracoid, the middle deltoid, the middle third of the scapula spine above and below and asking the patient to type of stimulus perceived (touch or pain).
Quantitative sensory testing (QST)-Mechanical allodynia | The outcome will be measured on day 1 for each site, by a physiotherapist during the clinical examination
  These tests will be adopted to assess peripheral and central sensitiazion phenomena. ests will be administered once for each site, by a physiotherapist using Neuropen.
  -Mechanical allodynia will be evaluated by maintaining the assessor's thumb with a standardized constant pressure for 10 seconds on the skin of middle deltoid, the anterior deltoid, the middle third of the scapular spine above and below, asking if the stimulus is painful.
Pain spatial summation to assess the pain descending inhibitory system | Tests will be administered on day 1 for each site, by a physiotherapist using Neuropen
  The wind-up phenomenon will be investigated by administering a set of 10 punctures on the skin of the middle deltoid, anterior deltoid, and middle third of the scapula above and below the scapula spine, asking if the patient to report initial and final pain rates through a Numeric Pain Rating Scale. The patient will be asked to give a verbal score on the pain intensity perceived. The score ranges from 0 (=no pain) to 10 (= maximum pain imaginable).

SECONDARY OUTCOMES:
International Classification of Functioning, Disability, and Health Generic Core Set | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to assess the subject's health status. It consists of 7 items and includes the following subcategories: body functions (physiological functions of the body system), body structures (anatomical components such as organs, limbs, and their components), activities (execution of a task or activity by an individual), and participation (involvement in daily life).
  Scale values are from 0 to 4 where 0 is the better outcome (no help needed) and 4 is the worse outcome (impossible to be performed alone)
Italian Shoulder Pain and Disability Index (SPADI-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to assess the disability of the upper limb. This scale consists of 13 items, which include two subcategories: 5 items assessing the pain-related disability and 8 items assessing the shoulder function. Scale values are from 0 to 130 where 0 is the better outcome (no disability) and 130 is the worse outcome (higher disability).
Italian Pain Catastrophizing Scale (PCS-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to assess the catastrophization. This scale consists of 13 items divided into three domains. Each item can achieve a maximum of 4 points, for a maximum of 52. The higher the score, the greater the presence of thoughts of catastrophization.
Italian Tampa Scale for Kinesophobia (TSK-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to measure kinesiophobia and fear of movement. This scale consists of 17 items assessing the fear of movement perception, scored 1 to 4 points (1=totally disagreeing: 4= strongly agree), achieving a score that varies between 17 and 68. The higher the score, the higher the level of fear related to movement.
Italian Hospital Anxiety Depression Scale (HADS-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to assess anxiety and depression.This scale consists of 14 items divided into two subcategories. The first 7 items investigate General anxiety, while the other 7 items, mainly investigate the state of anhedonia. For each item the score varies from 0-3 (0= absence; 3= extreme presence). Higher scores correspond to high levels of anxiety and depression.
Italian Pain Self-efficacy Questionnaire (PSEQ-I) | the self-reported scale will be administered on day 1, before the clinical examination
  It will be used to detect self-efficacy. This scale consists of 10 items, whose score varies from 0-6 (0=not safe at all, 10= completely safe), for a total of 60 points. The lower the score, the lower the self-efficacy is.
Upper Limb Neural Tension Test (ULNTT 1) | the test will be administered on day 1 by a physiotherapist during the clinical examination
  It will be used to assess mechanosensitivity of the brachial plexus and upper limb nerves. It consists of a validated combination of physiological movement of the arm (shoulder depression, wrist and finger extension, forearm supination, shoulder external rotation, and elbow extension) and a symptom discrimination maneuvers (homolateral and contralateral cervical spine inclination) to assess the physiological mechanosensitivity of the nerves of the upper limb.
Vagus nerve neurodynamic test (VN-NDT) | the test will be administered on day 1 by a physiotherapist during the clinical examination
  It will be performed to assess vagus nerve sensitization due to chronic stress. It consists of a combination of physiological movements of the neck (upper cervical flexion, contralateral lateral flexion, ipsilateral rotation) and gentle movements of the upper abdomen caudally and cranially to increase tension on the thoracic tract of the vagus nerve, and it assess the physiological mechanosensitivity of the vagus nerve and its effects on heart rate at rest.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Carta, MSc, PT BSc, Principal Investigator — University of Turin, Italy
Locations (1):
- Department of Biological and Clinical Science - University of Turin, Orbassano, TO, Italy

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available. All of the individual particiapnt data collected during the trial will be shared after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following the publication. No end date.
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.